CLINICAL TRIAL: NCT02443142
Title: Ibuprofen Versus Acetaminophen for Treatment of Mild Traumatic Brain Injury
Acronym: IVAMTBI
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of study participants.
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Demetrios Kyriacou, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NorthwesternU
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2015-03

CONDITIONS: Brain Concussion
Keywords: mild TBI; concussion; post-concussion syndrome
MeSH Terms: conditions — Brain Concussion; Post-Concussion Syndrome | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Experimental): Ibuprofen is a nonselective NSAID that inhibits both COX-1 and COX-2 isoenzymes. COX-2 inhibition prevents arachidonic acid from converting to vasoactive prostaglandins and reactive oxygen species in brain cell. The analgesic, antipyretic, and antiinflammatory activity of ibuprofen operates mainly through inhibition of COX-2. The experimental treatment oral doses of either ibuprofen (800 mg three times per day). Subjects will receive the first medication dose in the emergency department and will be given the remaining 5 doses to take over 48 hours as outpatients.
  Interventions: Drug: Ibuprofen
- Acetaminophen (Active Comparator): Acetaminophen is a poor inhibitor of both COX isoenzymes in the CNS and has significantly weaker antiinflammatory effects than NSAIDs. Acetaminophen does not inhibit COX in peripheral tissues and is less effective in the presence of peroxides. The active comparator treatment is oral doses of acetaminophen (1000 mg three times per day). Subjects will receive the first medication dose in the emergency department and will be given the remaining 5 doses to take over 48 hours as outpatients.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen 800 mg orally three times per day for two days for study subjects who are randomized to the ibuprofen arm.
  Other Names: motrin
  Arms: Ibuprofen
Drug: Acetaminophen — Acetaminophen 1000 mg orrally three times per day for two days for subjects who are randomized to the acetaminophen arm.
  Other Names: tylenol
  Arms: Acetaminophen

SUMMARY:
Traumatic brain injury (TBI) is an important public health problem with an estimated 1.7 million new cases in the United States each year. Although the vast majority of these victims sustain mild TBI, many still develop headache, difficulty concentrating, and decreased memory with potential for serious long-term consequences. In particular, mild TBI is an important consequence of combat-related injuries sustained by military personnel and sports-related injuries in young adults. Unfortunately, treatment of mild TBI is usually limited to oral analgesics for headache pain such as acetaminophen (Tylenol) or ibuprofen (Motrin or Advil). Since there are no previous randomized trials of these medications for mild TBI, their comparative effectiveness is not known. Increasing animal based evidence suggests that mild TBI is related to brain cell injury caused by overexpression of a cellular enzyme (COX-2) that causes neuroinflammation. Fortunately, inhibition of COX-2 is easily achieved using ibuprofen. We hypothesize that head injured patients treated with ibuprofen will have a lower incidence of mild TBI symptoms than patients treated with acetaminophen. We will conduct a randomized clinical trial to measure the comparative effects of ibuprofen versus acetaminophen on the incidence of specific symptoms of mild TBI in emergency department patients with head injury.

DETAILED DESCRIPTION:
OBJECTIVES

The long-term goal of the proposed project is to develop an effective pharmacological therapy for patients with mild TBI to improve functional outcomes. The main objective is to compare the effects of ibuprofen versus acetaminophen for reducing the short-term development post-concussion symptoms in patients with mild TBI. We will conduct a double-blinded randomized clinical trial (RCT) with the specific aim of measuring the comparative effects of equipotent doses of ibuprofen versus acetaminophen on the incidence of concussion symptoms to be measured 7 to 10 days after mild TBI in emergency department patients with isolated closed head injury. The main study hypothesis of our research project is that patients with mild TBI who are treated with ibuprofen will have a lower incidence of post-concussion symptoms compared to patients treated with acetaminophen. The proposed investigation is novel because it will be the very first RCT to compare analgesic medications for the specific treatment of mild TBI.

BACKGROUND

Pathophysiology of Mild TBI. TBI results from external mechanical force applied to the cranium leading to parenchymal brain damage. This resultant brain injury can range from mild temporary impairment to severe disability. TBI transpires in two phases: (1) primary brain injury occurs at the moment of the application of mechanical force on the cranium and results in lacerations, contusions, hematomas and shearing injuries of the brain; and (2) secondary brain injury begins immediately after the primary brain injury and results from the cellular mediation of neuroinflammation.15,16 The principal injury of mild TBI is diffuse axonal injury from shearing forces that is not usually identified by CT brain scan.17-20 Secondary brain injury activates multiple cellular pathways that are initially adaptive, but become pathological with overexpression and persistence.21-23 The biochemical consequences of these responses develop over a period of hours with the accumulation of arachidonic acid from cellular membrane stores and the induction of cyclooxygenase-2 (COX-2) gene expression and enzyme activity.15,16 Arachidonic acid is then converted to detrimental vasoactive prostanglandins and free radicals by COX-2 enzyme leading to neuronal cell death (Figure 1 see appendix). Neural COX-2 enzyme activity remains elevated for 1 to 3 days.24 Severity of neuronal injury is correlated to COX-2 overexpression which results in a "vicious cycle" of neuroinflammation when secondary injury propagates further COX-2 activity.15,16

Potential Effect of COX-2 Inhibition. If COX-2 overexpression causes neuronal cell damage after brain injury, then COX-2 inhibition may provide neuroprotective effects through two important mechanisms: (1) by reducing detrimental vasoactive prostanglandins and free radical synthesis; and (2) shunting of arachidonic acid down alternate pathways that produce beneficial eicosanoids.15 These cellular mechanisms are based on findings from several animal studies over the past 30 years that strongly suggest potential beneficial effects of NSAID inhibition of the COX-2 enzyme as a treatment for TBI-activated neuroinflammation.25-35 Although these studies examined different NSAID COX-2 kinhibitors and utilized different animal models of TBI, they found an overall consensus of beneficial effects (i.e., reduced prostaglandin synthesis, reduced brain edema, improvement in cognitive and motor function, improvements in memory, and reduced mortality) suggesting COX-2 inhibition may have effects beyond analgesia in patients with mild TBI. In fact, COX-2 inhibition has been shown to be beneficial for animal models for other types of brain insults including ischemic brain injury.36-40

If we identify a beneficial effect of ibuprofen for patients with mild TBI that is confirmed with validation studies, then new standards and guidelines will be developed to improve the ED management of this common form of brain injury. Future studies will be conducted to elaborate the effects of ibuprofen and other NSAIDS on both the short-term and long-term complications of mild TBI and possible other forms of TBI. Discovery of a beneficial effect of NSAIDs for mild TBI could be especially useful for combat-related and sports-related brain injuries.

STUDY DESIGN

Study subjects will be identified and enrolled in the emergency department. They will be followed for a 7 to 14 day period only. The proposed project will be completed over a one-year period with tasks and milestones as follows: Month 1 - develop protocol, create data collection instrument and codebook, test and modify instrument, create electronic database, and train assistants; Months 2 and 10 - identify and enroll eligible study subjects in the ED setting, create database, enter and edit data; and Months 11 and 12 - analyze data and interpret findings, prepare and submit papers to journals.

Study Design and Participants. We will conduct a double-blinded RCT to compare the effects of ibuprofen versus acetaminophen on the incidence of post-concussion symptoms measured 7 to 14 days after mild TBI.

Treatment Variable. The treatment variable will be equipotent oral doses of either ibuprofen (800 mg TID) or acetaminophen (1000 mg TID). Ibuprofen is a nonselective NSAID that inhibits both COX-1 and COX-2 isoenzymes. COX-2 inhibition prevents arachidonic acid from converting to vasoactive prostaglandins and reactive oxygen species in brain cell. The analgesic, antipyretic, and antiinflammatory activity of ibuprofen operates mainly through inhibition of COX-2.55,56 Acetaminophen is a poor inhibitor of both COX isoenzymes in the CNS and has significantly weaker antiinflammatory effects than NSAIDs. Acetaminophen does not inhibit COX in peripheral tissues and is less effective in the presence of peroxides.57,58 Both ibuprofen and acetaminophen are frequently prescribed for headache pain related to mild TBI in the ED and other primary care settings and have excellent safety profiles for short-term use. In fact, both ibuprofen and acetaminophen have been used for the antipyretic treatment of children with severe traumatic brain injury.59 Subjects will receive the first medication dose in the ED and will be given the remaining 5 doses to take over 48 hours as outpatients. This time period was selected based on animal models identifying maximum COX-2 activity. Both medications will be identically prepared to prevent subjects from identifying the type of treatment regimen. Treatment assignment will be randomized by the NMH research pharmacy and blinded to both the patients and the investigators. Standard methods for blinding will be implemented by using tablets that are identical in size, shape, color and taste for both ibuprofen and acetaminophen.

Data Collection and Variable Measurement. Information concerning the outcome and secondary study variables will be obtained by research assistants using standardized data collection instruments. Follow up outcome assessment will be conducted through telephone interviews at 7 to 14 days after head injury. We will implement best practice methods for accurate and complete data collection, including the following: (1) training assistants in data collection methods; (2) blinding assistants to the subjects' treatment assignment; and (3) conducting meetings with assistants to review data collection processes and difficulties. Subjects with persistent mild TBI symptoms at time of follow up will be referred to the Rehabilitation Institute of Chicago Concussion Clinic for further treatment.

Research Location. Northwestern Memorial Hospital is a state-of-the art, two million square foot, 873-bed tertiary teaching hospital in downtown Chicago that is the primary teaching hospital affiliated with the Northwestern University Feinberg School of Medicine. The Northwestern Memorial Hospital Emergency Department is an urban, academic, 56 bed, Level I trauma center with an annual patient volume of over 85,000 patients per year or approximately 230 patients per day. The Emergency Department is staffed exclusively by board-certified emergency medicine physicians that also supervise the care of 48 residents and four fellows. The reported demographic distribution of the overall Emergency Department patient population is as follows: 7% Hispanic; 2% Asian; 35% Black; and 63% White.

SATATISTICAL ANALYSES

Data Analyses Plan. We will conduct all statistical analyses based on the American Statistical Association Ethical Guidelines for Statistical Practice67,68 and include the following:

1. Univariate Analyses. We will first conduct univariate analyses to assess potential demographic and clinical differences between the two treatment groups. We will also use ANOVA to compare the effects of ibuprofen versus acetaminophen treatment on the incidence of mild TBI symptoms using continuous measures of pain scores and Neural-QOL measures of pain and cognitive function.
2. Multivariate Analyses. We will use log binomial regression modeling to adjust for potential residual confounding to estimate the effects of ibuprofen versus acetaminophen on the incidence of mild TBI symptoms. We will also conduct survival analyses using Kaplan-Meier graphs and Cox proportional hazards regression modeling to estimate adjusted hazards ratios for the effects of ibuprofen versus acetaminophen on the main outcomes of mild TBI symptoms. We will also conduct likelihood ratio and goodness-of-fit tests to identify and include specific covariates for the regression models and diagnostic methods to evaluate overall model fit and plausibility of model assumptions.
3. Advanced Methods for Causal Inference. We will use advanced statistical methods to allow assessment of causation: (1) instrumental variables to estimate the effects of ibuprofen versus acetaminophen with potential treatment regimen noncompliance by using treatment randomization as a perfect instrument;69,70 (2) marginal structural modeling to account for time-varying confounders and to assess for direct versus indirect effects in the presence of intermediate factors.71-74

Sample Size Estimation. Sample size estimation is especially challenging because there are no prior human studies measuring the effect of COX-2 inhibition on the incidence of mild TBI symptoms. Notwithstanding this limitation, we will use the presence of headache pain at 7 to 14 days as a binary outcome. Sample size estimation is based on the following: (1) 40% expected frequency of headache pain in the ibuprofen group versus 60% expected frequency in the acetaminophen group; (2) the use of two-sided tests performed at a significance level of 0.05; (3) a power of 0.80 to detect a true difference in headache pain between subjects receiving ibuprofen versus acetaminophen; and (4) one to one distribution of study subjects receiving ibuprofen versus acetaminophen. With these assumptions, the estimated number of study subjects needed to statistically assess ibuprofen versus acetaminophen for the treatment of mild TBI is a total of 214 subjects.60 Our plan to enroll over 400 subjects will provide an adequate sample size to conduct our statistical analyses. The Northwestern Memorial Hospital Emergency Department provides care to about 2,000 head injured patients with mild TBI each year.

ELIGIBILITY:
Inclusion Criteria:

1. Closed head injury within the past 24 hours with history (loss of consciousness, amnesia, mechanism of injury such as motor vehicle collision or fall from height) or specific symptoms and signs (headache, vomiting, dizziness, head injury, short-term memory deficit, confusion, blurred vision, balance problems) that prompts computerized tomography (CT) brain evaluation as determined by an emergency physician.
2. Age 21 through 60 years of age.
3. Initial Glasgow Coma Score of 13 or greater at time of ED presentation with normal neurologic examination and Glasgow Coma Score of 15 within two hours of initial assessment.
4. Normal neurologic examination in the emergency department except for symptoms and signs described above (e.g., no focal neurologic deficit).
5. Normal brain and skull on CT scan in the ED.
6. Working cellular phone (for follow up assessment).

Exclusion Criteria:

1. Significant concomitant non-cranial injury requiring pain medication (e.g., facial fracture, severe extremity injury, major blunt trauma.)
2. Any type of skull or cervical spine fracture.
3. Post-traumatic seizure.
4. Currently taking NSAIDS, acetaminophen, or other pain medications on a regular basis.
5. Currently taking ANY coagulant medication (e.g., Plavix, aspirin, Xeralto, Coumadin).
6. Any bleeding disorder, predisposition to bleeding, or history of gastrointestinal bleeding.
7. Pregnancy.
8. Clinical intoxication with alcohol or illicit medication.
9. Chronic alcohol abuse.
10. Any liver or renal dysfunction or failure.
11. Justification of obtaining CT brain evaluation that included patient being intoxicated.
12. Intolerance, allergy or adverse reaction to either ibuprofen or acetaminophen.
13. Any current or previously diagnosed cardiovascular condition (e.g., hypertension, coronary arterial disease, myocardial infarct, angina, congestive heart failure, pulmonary embolism, deep venous thrombosis).
14. Any current or previously diagnosed neurovascular condition (e.g., stroke, TIA, multiple sclerosis, seizure disorder).
15. Any active cancer or malignancy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05-01; Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Post-concussion symptoms | 7 to 14 days after enrollment.
  The main outcome variables will be the incidence of post-concussion symptoms that will be measured using NIH Common Data Elements and Neuro-QOL instruments. The Neuro-QOL instruments were developed for the NIH by the Northwestern University Department of Medical Social Sciences to provide clinically relevant and psychometrically robust health-related quality of life assessment tools for patients with common neurological disorders. In addition, the Neuro-QOL measurement system provides item banks and short forms that enable patient reported outcome measurement in neurological research which minimizes patient burden.41-44 This information will be collected at 7 to 14 days after initial ED evaluation. Emphasis will be placed on the Neuro-QOL instruments that measure headache pain and cognitive function as these are the most common and concerning symptoms of mild TBI.

SECONDARY OUTCOMES:
Adverse drug reactions | 7 to 14 days after enrollment
  Information regarding adverse drug reactions (ADRs) will also be obtained during the follow up interview of the study subjects. This assessment will include questions regarding abdominal pain or discomfort and any allergic reaction (e.g., rash, swelling, or difficulty breathing).

CONTACTS AND LOCATIONS:
Overall Officials: Demetrios N. Kyriacou, MD,PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States